CLINICAL TRIAL: NCT03546777
Title: Should the Coroacromial Ligament be Evaluated in Shoulder Magnetic Resonance Imaging?
Brief Title: Evaluation Coroacromial Ligament Thickness
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Çiğdem Aydoğan, Medical Doctor in Physical Medicine and Rehabilitation Clinic, Suleyman Demirel University
Other Study IDs: 37
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain, coracoacromial ligament thickness
MeSH Terms: conditions — Shoulder Pain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: magnetic resonance imaging — magnetic resonance imaging of shoulder

SUMMARY:
In this study, it was aimed to determine the relationship between pathologic findings and coracoacromial ligament thickness in magnetic resonance imaging in shoulder pain patients.

DETAILED DESCRIPTION:
The coracoacromial ligament, which is part of the coracoacromial arch, plays an important role in shoulder biomechanics, joint stability and proprioception. Age-related changes due to chronic stress and cellular impairment may contribute to thickening and stiffening of the coracoacromial ligament to rupture the rotator cuff and development of shoulder pathologies such as impingement syndrome. In this study, it was aimed to determine the relationship between pathologic findings and coracoacromial ligament thickness in magnetic resonance imaging in shoulder pain patients. Secondary purpose is whether the thickness of the coracoacromial ligament is indicative of shoulder pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 15 years diagnosed with shoulder pain

Exclusion Criteria:

* Sensation and reflexes loss in the upper extremity
* Limitation in passive shoulder movements on physical examination
* Systemic rheumatic disease
* Diabetes mellitus
* Malignant disease
* Active infection
* Intraarticular injection
* Trauma
* History of surgery

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with shoulder pain
Sampling Method: Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Thickness of coracoacromial ligament | 1 week
  magnetic resonance imaging of coracoacromial ligament

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Aydoğan, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided